CLINICAL TRIAL: NCT01365065
Title: A Pilot Study to Assess the Safety and Effect on HIV Transcription of Vorinostat in Patients Receiving Suppressive Combination Anti-retroviral Therapy
Brief Title: Safety and Effect on HIV Transcription of Vorinostat in Patients Receiving Suppressive Combination Anti-retroviral Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1121-9077
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: HIV Positive
MeSH Terms: conditions — HIV Seropositivity | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat (Experimental): Vorinostat 400mg ( 4 X 100mg ) orally daily for 14 days
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — Vorinostat 400mg (4 x 100mg) orally daily for 14 days

SUMMARY:
The objective of the study is to assess the safety and ability of vorinostat, a drug currently licensed for the treatment of a type of lymphoma, to 'turn on' dormant HIV infected CD4 T-cells.

DETAILED DESCRIPTION:
Treatment of HIV infection with combination antiretroviral therapy (cART) has led to significant improvements in the life expectancy and quality of life of people living with HIV. Nevertheless, life expectancy is significantly lower than uninfected individuals and cART leads to several long term side effects. cART alone is not able to cure HIV infection due to persistence of HIV infection in dormant cells. One potential strategy to eradicate HIV infection is to 'wake up' these dormant infected cells by 'turning on' the cell. The small number of cells that are dormant and infected would start to produce virus and die, but infection of other cells would be prevented by cART. Ultimately this could lead to eradication of dormant infected cells and a potential cure for HIV.

This study is a pilot study in 20 individuals recruited at the Alfred Hospital only.

The hypotheses is that vorinostat will induce HIV transcription in CD4 T-cells with latent HIV infection, it is safe and well tolerated in patients receiving effective cART and will induce histone acetylation in vivo in patients with HIV infection.

The study will run over 12 weeks, involving 9 study visits for the participant. Eligible patients must be between 18 to 60 years of age with confirmed HIV infection, and receiving successful cART as indicated by 'suppressed' HIV virus in blood (plasma HIV RNA <50 copies/ml) for at least 3 years and a strong immune system (two CD4 counts greater than 500 cell/µl in the last 6 months).

Patients will be reviewed at screening and days 1 (three time points), 2, 7, 14, 21, 28 and 84 (week 12). They will have blood tests for HIV viral load assessment, CD4 cell counts, biochemistry, hematology and storage samples. An electrocardiogram of the heart (ECG) will be taken at screening, day 7 and 14.

As part of this study levels of HIV in blood and in white blood cells and the degree to which cells are 'turned on' (histone (H3) acetylation) will be measured at 3 time points on day 1, then once on days 2, 7, 14, 21 and 28. The level of one component of cART will be measured at day 1 and 14. At baseline and day 14 a sigmoidoscopy if performed for the collection of rectal biopsies.

The safety and how well vorinostat is tolerated will be determined based on physical exams, laboratory tests and questions about any problems patients may have experienced during the study. This study has an Independent Safety Monitoring Committee who in addition to evaluating the overall safety of patients will be responsible for assessing safety of the first patient enrolled prior to any recommendation to continue the study.

ELIGIBILITY:
Inclusion Criteria:

1. HIV -1 infected adults
2. HIV-1 plasma RNA <50 copies/ml for at least 3 years with at least 2 viral load measures per year, and most recent viral load within 3 months of screening. Episodes of a single HIV plasma RNA 50-199 copies/ml will not exclude participation if the subsequent HIV plasma RNA was <50 copies/ml.
3. Receiving combination antiretroviral therapy (at least 3 agents)
4. In the last 6 months have two CD4 cell count greater than 500 cell/µl
5. Documented subtype B HIV infection
6. Detectable HIV RNA on stored specimen
7. Able to give informed consent

Exclusion Criteria:

1. Any significant acute medical illness in the past 8 weeks.
2. Any evidence of an active AIDS-defining opportunistic infection.
3. Current or recent gastrointestinal disease that may impact the absorption of study drug.
4. Any gastrointestinal surgery that could impact upon the absorption of study drug.
5. Active alcohol or substance use that, in the Investigator's opinion, will prevent adequate compliance with study therapy .
6. Moderate to severe hepatic impairment
7. Hepatic transaminases (AST or ALT) > 3 x upper limit of normal (ULN)
8. Hepatitis B infection as indicated by the presence of Hepatitis B surface antigen or detectable DNA levels in blood.
9. A personal history of clinically significant cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de pointes (e.g. heart failure).
10. History of malignancy or transplantation, including skin cancers or Kaposi sarcoma
11. History of diabetes mellitus
12. Use of an HIV protease inhibitor.
13. Receipt of immunomodulating agents, immunization or systemic chemotherapeutic agents within 28 days prior to screening.
14. Use of an agent definitely or possibly associated with effects on QT intervals within 2 weeks of screening.
15. Receipt of sodium valproate or other HDAC inhibitor at any time.
16. Women who are pregnant or breastfeeding, or with a positive pregnancy test during screening or Women of Child Bearing Potential (WOCBP) who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for the entire study period and for at least 4 weeks before and 4 weeks after the study.
17. Males who are unwilling or unable to use barrier contraception during vaginal intercourse from the time of enrollment and for 12 weeks after participation in the study are also excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of vorinostat on HIV transcription in CD4 T-cells. | Day 1 (before drug, 2 and 8 hours after first dose), Day 2, 7, 14, 21 and 28
  The primary (efficacy) endpoint of this study is to evaluate the effect of vorinostat on HIV transcription from latently infected CD4+ T-cells as measured by HIV unspliced RNA in CD4+ T-cells.

SECONDARY OUTCOMES:
1. To evaluate the safety and tolerability of vorinostat in patients receiving effective combination antiretroviral therapy (cART | Screening, Day 1, 7, 14,21, and 28
  1. Plasma HIV RNA (standard assay)
  2. Adverse events and dose-limiting toxicity
  3. CD4 T-cell count
  4. Antiretroviral plasma trough concentrations will be measured before and after 14 days of treatment with vorinostat.

CONTACTS AND LOCATIONS:
Locations (1):
- The Alfred Hospital - Infectious Diseases Unit, Melbourne, Victoria, Australia

REFERENCES:
- [Result] Elliott JH, Wightman F, Solomon A, Ghneim K, Ahlers J, Cameron MJ, Smith MZ, Spelman T, McMahon J, Velayudham P, Brown G, Roney J, Watson J, Prince MH, Hoy JF, Chomont N, Fromentin R, Procopio FA, Zeidan J, Palmer S, Odevall L, Johnstone RW, Martin BP, Sinclair E, Deeks SG, Hazuda DJ, Cameron PU, Sekaly RP, Lewin SR. Activation of HIV transcription with short-course vorinostat in HIV-infected patients on suppressive antiretroviral therapy. PLoS Pathog. 2014 Nov 13;10(10):e1004473. doi: 10.1371/journal.ppat.1004473. eCollection 2014 Oct. PMID 25393648
- [Result] Mota TM, Rasmussen TA, Rhodes A, Tennakoon S, Dantanarayana A, Wightman F, Hagenauer M, Roney J, Spelman T, Purcell DFJ, McMahon J, Hoy JF, Prince HM, Elliott JH, Lewin SR. No adverse safety or virological changes 2 years following vorinostat in HIV-infected individuals on antiretroviral therapy. AIDS. 2017 May 15;31(8):1137-1141. doi: 10.1097/QAD.0000000000001442. PMID 28301423